CLINICAL TRIAL: NCT01323621
Title: A 12-week Study to Evaluate the 24-hour Pulmonary Function Profile of Fluticasone Furoate/Vilanterol (FF/VI) Inhalation Powder 100/25 mcg Once Daily Compared With Fluticasone Propionate/Salmeterol Inhalation Powder 250/50 mcg Twice Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study Evaluating the 24-Hour Pulmonary Function Profile of Fluticasone Furoate (FF) /GW642444 (Vilanterol) (VI) Inhalation Powder 100/25mcg Once Daily Compared With Fluticasone Propionate/Salmeterol Inhalation Powder 250/50mcg Twice Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112352
Record Dates: First submitted 2011-03-17; First posted 2011-03-25 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol; Fluticasone; Salmeterol Xinafoate; Albuterol; Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate / GW642444 (vilanterol) (Experimental): Inhaled Corticosteroid (ICS)/ Long acting Beta Agonist (LABA)
  Interventions: Drug: Fluticasone Furoate 100mcg/ GW642444 (vilanterol) 25mcg; Drug: Double-dummy placebo; Drug: Salbutamol as needed
- Fluticasone Propionate / salmeterol (Active Comparator): Inhaled Corticosteroid (ICS)/ Long acting Beta Agonist (LABA)
  Interventions: Drug: Fluticasone Propionate 250mcg / salmeterol 50mcg; Drug: Double-dummy placebo; Drug: Salbutamol as needed

INTERVENTIONS:
Drug: Fluticasone Furoate 100mcg/ GW642444 (vilanterol) 25mcg — inhalation powder
  Arms: Fluticasone Furoate / GW642444 (vilanterol)
Drug: Fluticasone Propionate 250mcg / salmeterol 50mcg — inhalation powder
  Arms: Fluticasone Propionate / salmeterol
Drug: Double-dummy placebo — inhalation powder
Drug: Salbutamol as needed — inhalation powder

SUMMARY:
The purpose of this study is to evaluate the 24-hour spirometry effect (FEV1) of FF/VI 100/25mcg once daily compared with Fluticasone Propionate/Salmeterol 250/50mcg twice daily over a 12-week treatment period in subjects with COPD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, multi-centre parallel group study. Subjects who meet the eligibility criteria at Screening and meet the randomization criteria at the end of a 2-week Run-In period will enter a 12-week treatment period. There will be a 7-day Follow-up period after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Male or females ≥ 40 years of age
* Established clinical history of COPD by ATS/ERS definition
* Females are eligible to enter and participate if of non-childbearing potential, or if of child bearing potential, has a negative serum pregnancy test at screening, and agrees to one of the acceptable contraceptive methods listed in protocol, used consistently and correctly
* Former or current smoker > 10 pack years
* Post-albuterol spirometry criteria: FEV1/FVC ratio ≤ 0.70 and FEV1 ≤ 70% of predicted normal (NHANES III)

Exclusion Criteria:

* Current diagnosis of asthma
* Subjects with other respiratory disorders including active tuberculosis, α1-antitrypsin deficiency, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Lung volume reduction surgery within previous 12 months
* Clinically significant abnormalities not due to COPD by chest x-ray
* Hospitalized for poorly controlled COPD within 12 weeks of Screening
* Poorly controlled COPD 6 weeks prior to Screening, defined as acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician
* Lower respiratory infection requiring antibiotics 6 weeks prior to Screening
* Uncontrolled or clinically significant (in opinion of PI) cardiovascular, hypertension, neurological, psychiatric, renal, hepatic, immunological, endocrine, peptic ulcer disease, or hematological abnormalities
* Carcinoma not in complete remission for at least 5 years
* Subjects with history of hypersensitivity to study medications (e.g., beta-agonists, corticosteroid) or components of inhalation powder (e.g., lactose, magnesium stearate)
* Subjects with history of severe milk protein allergy that, in opinion of study physician, contraindicates subject's participation
* Known/suspected history of alcohol or drug abuse in the last 2 years
* Women who are pregnant or lactating or plan to become pregnant
* Subjects medically unable to withhold albuterol and/or ipratropium 4 hours prior to spirometry testing at each study visit
* Use of certain medications such as bronchodilators and corticosteroids for the protocol-specific times prior to Visit 1 (the Investigator will discuss the specific medications)
* Long Term Oxygen Therapy (LTOT) or nocturnal oxygen therapy >12 hours a day
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening or during the study
* Non-compliance or inability to comply with study procedures or scheduled visits
* Affiliation with investigator site

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2011-03-18; Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (13):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Boerne, Texas
- GSK Investigational Site, Lübeck, Schleswig-Holstein, Germany
- Italy (11):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, San Felice A Cancello Caserta, Campania
  - GSK Investigational Site, Telese Terme (BN), Campania
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Torrette (AN), The Marches
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto
- South Africa (10):
  - GSK Investigational Site, Benoni, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, George
  - GSK Investigational Site, Port Elizabeth
  - GSK Investigational Site, Reiger Park
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Thabazimbi
  - GSK Investigational Site, Witbank
- Spain (6):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Lugo
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Valladolid
- Ukraine (7):
  - GSK Investigational Site, Cherkassy
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Dransfield MT, Feldman G, Korenblat P, LaForce CF, Locantore N, Pistolesi M, Watkins ML, Crim C, Martinez FJ. Efficacy and safety of once-daily fluticasone furoate/vilanterol (100/25 mcg) versus twice-daily fluticasone propionate/salmeterol (250/50 mcg) in COPD patients. Respir Med. 2014 Aug;108(8):1171-9. doi: 10.1016/j.rmed.2014.05.008. Epub 2014 Jun 19. PMID 24998880
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112352 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112352 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112352 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112352 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112352 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112352 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112352 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Visit 1, eligible participants entered a 2-week, single blind (placebo) Run-In Period to obtain Baseline assessments of albuterol (salbutamol) use and to evaluate adherence with study treatment and procedures, diary card completion, and assessment of disease stability. At Visit 2, participants were randomized to a 12-week Treatment Period.
Groups:
- Placebo + Salbutamol: Participants were instructed to take single-blind placebo (ACCUHALER/DISKUS and Novel Dry Powder Inhaler [NDPI]): one inhalation each morning from each device, and one inhalation from the ACCUHALER/DISKUS in the evening. In addition, all participants received supplemental albuterol (salbutamol) (metered dose inhaler [MDI] and/or nebules) to be used on an as-needed basis. Ipratropium bromide alone was permitted, provided that the participant was on a stable dose from Visit 1 (Screening) and remained on the stable dose throughout the study; however, Ipratropium must have been withheld for 4 hours prior to and during each clinic visit.
- FSC 250/50 µg BID: Participants received a Fluticasone Propionate and Salmeterol (FSC) 250/50 microgram (µg) inhalation (available as a combination dry inhalation powder of Fluticasone 250 µg and Salmeterol 50 µg in a single strip) twice daily (BID) (morning and evening) from the ACCUHALER/DISKUS and placebo once daily (QD) in the morning from the NDPI over the course of 12 weeks.
- FF/VI 100/25 µg QD: Participants received a Fluticasone Furoate /Vilanterol (FF/VI) 100/25 µg inhalation (available as a dry inhalation powder in two separate strips of FF 100 µg and VI 25 µg) QD in the morning from the NDPI and placebo BID (morning and evening) from the ACCUHALER/DISKUS over the course of 12 weeks.
Period: 2-week, Single-blind Run In Period
Arm/Group | Placebo + Salbutamol | FSC 250/50 µg BID | FF/VI 100/25 µg QD
Started | 739 | 0 | 0
Completed | 511 | 0 | 0
Not Completed | 228 | 0 | 0
Not completed — Not Met Inclusion/Exclusion Criteria | 121 | 0 | 0
Not completed — Physician Decision | 7 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 86 | 0 | 0
Period: 12-week, Double-blind Treatment Period
Arm/Group | Placebo + Salbutamol | FSC 250/50 µg BID | FF/VI 100/25 µg QD
Started | 0 | 252 | 259
Completed | 0 | 237 | 239
Not Completed | 0 | 15 | 20
Not completed — Adverse Event | 0 | 1 | 5
Not completed — Lack of Efficacy | 0 | 2 | 6
Not completed — Protocol Violation | 0 | 4 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSC 250/50 µg BID | FF/VI 100/25 µg QD | Total
Number analyzed (Participants) | 252 | 259 | 511
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (9.05) | 61.6 (9.59) | 61.6 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 78 | 163
  Male | 167 | 181 | 348
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European Heritage | 238 | 241 | 479
  African American/African Heritage | 14 | 17 | 31
  White - Arabic/North African Heritage | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Trough in 24-Hour Weighted Mean FEV1 on Treatment Day 84
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean was calculated from the pre-dose FEV1 and the post-dose FEV1 measurements at 5, 15, 30, and 60 minutes (min) and 2, 4, 6, 8, 12, 13, 14, 16, 20, and 24 hours post-dose on Treatment Day 84. Baseline trough FEV1 was calculated as the mean of the two assessments made 30 and 5 minutes pre-dose on Treatment Day 1. Change from Baseline was calculated as the average of the Day 84 values minus the Baseline value. Analysis of covariance (ANCOVA) was conducted with covariates for country, smoking status, reversibility, and Baseline FEV1.
Time Frame: Baseline (Day 1) and Day 84
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study drug. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FSC 250/50 µg BID | FF/VI 100/25 µg QD
Number analyzed (Participants) | 217 | 219
Liters | 0.114 (0.0183) | 0.142 (0.0182)
Statistical Analysis 1: Comparison: FSC 250/50 µg BID vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p = 0.267, ANCOVA; Least squares mean difference = 0.029, 95% CI [-0.022 to 0.080] — ANCOVA analysis was conducted with covariates for country, smoking status, reversibility, and Baseline FEV1

2. Secondary Outcome: Time to Onset on Treatment Day 1
Description: Time to onset on Treatment Day 1 is defined as the time to an increase of 100 milliliters (mL) from Baseline in FEV1. Time to onset was calculated over 0 to 4 hours (5 min, 15 min, 30 min, 60 min, 120 min, and 240 min) post-dose.
Time Frame: Baseline and Day 1
Population: ITT Population
Measure: Median (Full Range); unit: Minutes
Arm/Group | FSC 250/50 µg BID | FF/VI 100/25 µg QD
Number analyzed (Participants) | 251 | 258
Minutes | 30 [5 to 240] | 16 [5 to 240]

ADVERSE EVENTS:
Arm/Group | FSC 250/50 µg BID | FF/VI 100/25 µg QD
Serious Adverse Events (participants affected / at risk) | 3/252 | 5/259
Other Adverse Events (participants affected / at risk) | 10/252 | 12/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC 250/50 µg BID (N=252) | FF/VI 100/25 µg QD (N=259)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FSC 250/50 µg BID (N=252) | FF/VI 100/25 µg QD (N=259)
Headache (Nervous system disorders) | 10 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.